CLINICAL TRIAL: NCT05031416
Title: Developing and Pilot Testing a Remote Smoking Cessation Digital Therapeutic for Individuals With Serious Mental Illness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to proceed with the study at this time.
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00273925; P50MH115842 (NIH)
Record Dates: First submitted 2021-08-12; First posted 2021-09-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consumers who smoke at outpatient community mental health clinic (Experimental): Consumers with serious mental illness who attend outpatient community mental health clinic will participate in a smoking cessation with the LTQ application and nicotine replacement therapy
  Interventions: Combination Product: LTQ

INTERVENTIONS:
Combination Product: LTQ — The investigators will test the LTQ-Connect application and a standard 10-week course of nicotine replacement therapy (NRT) nicotine patches, and Facebook groups, which will run for a total of 3 months with research study participants

SUMMARY:
This is a pilot randomized clinical trial testing an implementation intervention to support delivery of a smoking cessation app tailored to the needs of those individuals with SMI who at community mental health programs.

DETAILED DESCRIPTION:
Learn to Quit (LTQ), an evidence-based smoking cessation app tailored to the needs of individuals with serious mental illness (SMI) that demonstrated promising smoking cessation outcomes in a recent pilot randomized controlled trial (R00 DA037276). In parallel, several trials demonstrated that widely available social media platforms can be effectively utilized to enhance the effects of standard of care evidence-based smoking cessation treatments. Both approaches capitalize on highly scalable digital technologies, and are therefore likely to have population level impact. Drawing from these two separate programs of research, the central premise of this proposal is that LTQ, a stand-alone smoking cessation app tailored to patients with SMI, can be enhanced with peer-support delivered on social media. Therefore, this proposal seeks to develop and asses the acceptability and feasibility of LTQ-Connect -- the integration of the evidence-based smoking cessation app, LTQ, with social support delivered via social media -- to boost the efficacy and community reach of digital therapeutics tailored for patients with SMI. To achieve this goal, we will:

(1) determine the ideal design requirements of an LTQ-Connect integration among smokers with SMI, and (2) investigate the feasibility of LTQ-Connect in a single group pilot trial. Both interventions will be combined with nicotine replacement therapy, a safe and widely available medication.

ELIGIBILITY:
Inclusion Criteria:

* Must be a mental health consumer at Johns Hopkins Bayview Adult Psychiatry Program
* A regular smoker who is willing to quit
* Own a smart cell phone
* Willing to participate

Exclusion Criteria:

* Women who report being pregnant or have the intention to become pregnant in the 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Self reported social support | 13 weeks
  An adapted version of Online Social Support (OSS) scale for smokers will be used to evaluate self-reported social support from online smoking cessation treatment (LTQapp + Facebook group) The OSS scale is a 14 item scale with choices - 1 disagree a lot, to 4 agree a lot. Scale range 14- 56 with higher score indicating better outcome.
App Usability | 13 weeks
  The System Usability Scale (SUS) is a 10-item scale used to evaluate usability of the LTQ-Connect app. Choices range from 1 strongly disagree, to 5 Strongly agree. Scale range 10-50 with higher score indicating more agreement.
Number of user Interactions with the Learn to Quit (LTQ) app | 13 weeks
  Google Analytics will be used to extract number of daily app interactions and duration of engagement with LTQ app.
Duration of user Interactions with the Learn to Quit (LTQ) app | 13 weeks
  Google Analytics will be used to extract daily duration of interactions with LTQ app in minutes.
User Engagement with Facebook groups - Posts | 13 weeks
  The Facebook API will be used to extract number of Facebook posts.
User Engagement with Facebook groups - Comments | 13 weeks
  The Facebook application programming interface (API) will be used to extract number of Facebook comments.
User Engagement with Facebook groups - Likes | 13 weeks
  The Facebook API will be used to extract number of Facebook likes.
User Engagement with Facebook groups - Content | 13 weeks
  The Facebook API will be used to extract engagement content of Facebook posts, comments, and 'likes.'

SECONDARY OUTCOMES:
Change in number of cigarettes smoked per day | Week 5, Week 9, and Week 13
  The Smoking timeline follow-back (TLFB) will be used to estimate the number of cigarettes per day
Psychiatric Functioning | Week 5, Week 9, and Week 13
  The Brief Symptom Inventory (BSI) assesses distress participants are experiencing. The BSI is a 13 item scale with choices 0=not at all, to 4= Extremely. A higher score indicates more distress. Score range 0-52.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Daumit, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No